CLINICAL TRIAL: NCT06817239
Title: Effect of Perioperative Low-dose EsketaMine on dElirium in High-risk Elderly Patients uNdergoing elecTive Major Non-cardiac Surgery: a Multi-center Randomized Trial (ELEMENT Trial)
Brief Title: Effect of Low-dose EsketaMine on dElirium in High-risk Elderly Patients uNdergoing elecTive Surgery (ELEMENT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NFEC-2025-016
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Delirium in Old Age; Delirium, Postoperative; Anesthesia; Cognitive Dysfunction; Pain, Postoperative; Esketamine; Non-cardiac Surgery
Keywords: Delirium; Elderly patients; Esketamine; Non-cardiac surgery
MeSH Terms: conditions — Emergence Delirium; Cognitive Dysfunction; Pain, Postoperative; Delirium | interventions — Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine (Experimental): Esketamine (1mg/ml) will be administered at a loading dose of 0.2 mg/kg, namely at a infusion rate of 1.2ml/kg/h over 10 minutes after induction, then a maintenance infusion rate of 0.1 mg/kg/h until 40 minutes before the end of the surgery. For postoperative analgesia, patient-controlled intravenous analgesia (PCIA) is prepared with a formulation consisting of esketamine 50mg and sufentanil 200 μg, diluted to a total volume of 200 ml. The background dose is set at 2 ml/h, with a bolus dose of 2 ml and a lockout interval of 15 minutes.
  Interventions: Drug: Esketamine
- Normal saline (Placebo Comparator): Normal saline will be administered at a infusion rate of 1.2ml/kg/h over 10 minutes after induction, then a maintenance infusion rate of 0.1 mg/kg/h until 40 minutes before the end of the surgery. For postoperative analgesia, patient-controlled intravenous analgesia (PCIA) is prepared with sufentanil 200μg, diluted to a total volume of 200 ml. The background dose is set at 2 ml/h, with a bolus dose of 2 ml and a lockout interval of 15 minutes.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Esketamine — Esketamine (1mg/ml) will be administered at a loading dose of 0.2 mg/kg, namely at a infusion rate of 1.2ml/kg/h over 10 minutes after induction, then a maintenance infusion rate of 0.1 mg/kg/h until 40 minutes before the end of the surgery. For postoperative analgesia, patient-controlled intravenous analgesia (PCIA) is prepared with a formulation consisting of esketamine 50mg and sufentanil 200 μg, diluted to a total volume of 200 ml. The background dose is set at 2 ml/h, with a bolus dose of 2 ml and a lockout interval of 15 minutes.
  Arms: Esketamine
Drug: Normal saline — Normal saline will be administered at a infusion rate of 1.2ml/kg/h over 10 minutes after induction, then a maintenance infusion rate of 0.1 mg/kg/h until 40 minutes before the end of the surgery. For postoperative analgesia, patient-controlled intravenous analgesia (PCIA) is prepared with sufentanil 200μg, diluted to a total volume of 200 ml. The background dose is set at 2 ml/h, with a bolus dose of 2 ml and a lockout interval of 15 minutes.
  Arms: Normal saline

SUMMARY:
Delirium is an acutely occurred neurocognitive disorder characterized by fluctuating symptoms of inattention, altered consciousness and cognitive dysfunction. Delirium is reported to occur in 4% to 65% of postoperative patients depending on the population, and is especially common in older patients. Postoperative delirium is disturbing to patients and their families, and it is a strong predictor of both early and long-term worse outcomes including increased non-delirium complications, increased perioperative mortality, shortened overall survival, declined cognitive function, and lowered quality of life.

Although ketamine/esketamine has anti-inflammatory and neuroprotective effects, evidence on its efficacy in reducing postoperative delirium remains inconsistent and inconclusive. Existing studies are limited by heterogeneity, small sample sizes, single-center designs, and a focus on specific type of surgery. Research on elderly high-risk patients is lacking, and most studies administer the drug intraoperatively, with limited exploration of postoperative use. The optimal dosing and timing for POD prevention are unclear. This study aims to carry out a multicenter, single-blind, placebo-controlled, large-sample randomized controlled trial assessing the effect of low-dose esketamine, given intraoperatively and postoperatively, on delirium in elderly high-risk patients undergoing major non-cardiac surgery.

DETAILED DESCRIPTION:
Delirium is an acutely occurred neurocognitive disorder characterized by fluctuating symptoms of inattention, altered consciousness and cognitive dysfunction. Delirium is reported to occur in 4% to 65% of postoperative patients depending on the population, and is especially common in older patients. Postoperative delirium is disturbing to patients and their families, and it is a strong predictor of both early and long-term worse outcomes including increased non-delirium complications, increased perioperative mortality, shortened overall survival, declined cognitive function, and lowered quality of life.

The mechanism of delirium remains unclear, with neuroinflammation playing a significant role. Emerging evidence suggests anesthetic drug selection may influence the incidence of delirium. Ketamine, a non-competitive NMDA receptor antagonist, exhibits anti-inflammatory and neuroprotective properties by reducing TNF-α, IL-6, IL-1β, p-TAU, and S100B levels, mitigating oxidative stress, and inhibiting neuronal autophagy via the PI3K/AKT/mTOR pathway, thereby potentially preserving cognitive function. Clinical studies exploring ketamine's role in postoperative delirium have yielded mixed results. A retrospective study involving ICU patients undergone abdominal surgery found low-dose ketamine reduced delirium risk by 43% after propensity score matching. In cardiac surgery patients, a single dose of ketamine during induction decreased delirium incidence from 31% to 3%. However, a large international multicenter RCT in patients aged ≥60 undergoing major surgery found no reduction in delirium with pre-induction ketamine. A meta-analysis of eight RCTs also reported no preventive effect, though significant heterogeneity and inconsistent diagnostic criteria were noted. Perioperative ketamine use was consistently found safe, with no increase in adverse events such as nausea, vomiting, respiratory depression, or psychiatric symptoms.

Esketamine, the S-(+)-enantiomer of ketamine, has higher bioavailability, a shorter elimination half-life, and fewer side effects. It is effective in general anesthesia, postoperative analgesia, and ICU sedation, and can be used alone for minor procedures or combined with general or regional anesthesia. As an adjunct, it reduces the need for sedatives (e.g., propofol, midazolam) and opioids, minimizes hemodynamic fluctuations and respiratory depression, and improves anesthesia safety. Esketamine may prevent postoperative delirium, as suggested by emerging evidence. A single dose (0.25 mg/kg) before induction reduced delirium incidence in cardiac surgery patients from 44.6% to 23.2%. In elderly patients undergone gastrointestinal cancer surgery, intraoperative infusion (0.25 mg/kg at induction, then 0.125 mg/kg/h until 20 minutes before the end of surgery) decreased delayed neurocognitive recovery but not delirium. Conversely, postoperative esketamine (1 mg/kg) reduced delirium incidence from 40% to 13.3% in another RCT involving elderly patients undergone gastrointestinal surgery. In patients after major abdominal surgery, mini-dose esketamine (0.015 mg/kg/h for 48 hours) significantly lowered ICU delirium scores compared to low-dose esketamine or placebo. Two meta-analyses of 13 and 17 RCTs, respectively, reported reduced delirium incidence with perioperative esketamine usage, though evidence quality was limited by small sample sizes and heterogeneity. Recent studies showed mixed results. A single-center RCT of 426 elderly surgical patients found no reduction in delirium with 0.2 mg/kg esketamine at induction. In 209 patients aged ≥60 undergone tumor resection, 0.5 mg/kg at induction and 2 mg/kg PCIA postoperatively did not reduce delirium but may improve 90-day cognitive function. Similarly, a single-center RCT of 260 elderly patients after arthroplasty surgery found no benefit with esketamine administered at induction (0.2 mg/kg), intraoperatively (0.125 mg/kg/h), and postoperatively (0.5 mg/kg PCIA). Despite inconsistent findings, esketamine is safe in total, with no increased risk of adverse effects such as respiratory depression, nausea, vomiting, or psychiatric symptoms.

Although ketamine/esketamine has anti-inflammatory and neuroprotective effects, evidence on its efficacy in reducing postoperative delirium remains inconsistent and inconclusive. Existing studies are limited by heterogeneity, small sample sizes, single-center designs, and a focus on specific type of surgery. Research on elderly high-risk patients is lacking, and most studies administer the drug intraoperatively, with limited exploration of postoperative use. The optimal dosing and timing for POD prevention are unclear. This study aims to carry out a multicenter, single-blind, placebo-controlled, large-sample randomized controlled trial assessing the effect of low-dose esketamine, given intraoperatively and postoperatively, on delirium in elderly high-risk patients undergoing major non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years and <90 years;
* Scheduled to undergo major non-cardiac surgery.
* Fulfill at least one of risk factors as follows: history of stroke; history of delirium; hypertension; congestive heart failure; coronary artery disease; atrial fibrillation; peripheral artery disease; chronic obstructive pulmonary disease; obstructive sleep apnea; diabetes; chronic kidney disease; anemia; malnutrition; hypoalbuminemia; chronic pain; anxiety and depression; poor sleep quality; smoke; alcoholism.
* Scheduled to receive patient-controlled intravenous analgesia (PCIA).

Exclusion Criteria:

* Refuse to participate;
* Preoperative history of epilepsy, myasthenia gravis, Parkinson's disease, intracranial hypertension, delirium, schizophrenia, or other psychiatric diseases;
* Inability to communicate in the preoperative period because of coma, profound dementia, or language barrier;
* Preoperative uncontrolled severe hypertension (baseline SBP>180 mmHg or DBP>110 mmHg);
* Preoperative history of hyperthyroidism and pheochromocytoma;
* Acute cardiovascular event occurring within 30 days before surgery;
* Severe hepatic dysfunction (Child-Pugh class C), renal dysfunction (required preoperative dialysis), or expected survival ≤24 hours;
* Scheduled to undergo organ transplantation, vascular surgery, neurosurgery;
* Receiving treatment with ketamine or esketamine;
* Contradiction to ketamine or esketamine;
* Other situations where the investigator or physician considers the patient ineligible for the study.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1670 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of delirium within 5 days after surgery | Up to 5 days after surgery
  Delirium is assessed twice daily (8-10 am and 6-8 pm) with The Confusion Assessment Method (CAM) for non-intubated patients or The confusion assessment method for the Intensive Care Unit (CAM-ICU) for intubated patients.
Quality of recovery on postoperative day 1 (Sub-study) | On postoperative day 1
  Quality of recovery is assessed once daily (6-8 pm) with 15-item Quality of Recovery Scale (QoR-15).

SECONDARY OUTCOMES:
Intensity of pain during the first 3 postoperative days | Up to 3 days after surgery
  Intensity of pain will be assessed twice after surgery with the Behavioral Pain Scale and Numeric Rating Scale (an 11- point scale where 0 indicates no pain and 10 the worst pain).
Use of opioids during the first 3 postoperative days | Up to 3 days after surgery
  Include opioids used for PCIA and supplemental analgesics.
Cognitive function at 30 days after surgery | At the end of 30 days after surgery
  Cognitive function is assessed with the Telephone-Montreal Cognitive Assessment (T-MoCA) (a 22-point scale, with higher score indicating better function).
The incidence of delayed neurocognitive recovery | At the end of 30 days after surgery
  A decline in the T-MoCA score by 1 standard deviation (SD) or more from the baseline is considered delayed neurocognitive recovery.
Death rate at 30 days after surgery | At the end of 30 days after surgery
  Survival status is followed up at 30 days after surgery.
Quality of recovery on postoperative day 3 (Sub-study) | On postoperative day 3
  Quality of recovery is assessed once daily (6-8 pm) with QoR-15.
Postoperative gastrointestinal intolerance during the first 2 postoperative days (Sub-study) | Up to 2 days after surgery
  Gastrointestinal intolerance is assessed once daily (6-8 pm) with Intake, Feeling nauseated, Emesis, Exam, and Duration of symptoms scoring system (I-FEED).
Postoperative gastrointestinal dysfunction during the first 2 postoperative days (Sub-study) | Up to 2 days after surgery
  Gastrointestinal dysfunction is assessed once daily (6-8 pm) with Intake, Feeling nauseated, Emesis, Exam, and Duration of symptoms scoring system (I-FEED).
Quality of recovery at 30 days after surgery (Sub-study) | At the end of 30 days after surgery
  Quality of recovery is assessed with QoR-15.
HADS score at 30 days after surgery (Sub-study) | At the end of 30 days after surgery
  Anxiety and depression are assessed with Hospital Anxiety and Depression Scale (HADS).
Sleep quality at 30 days after surgery (Sub-study) | At the end of 30 days after surgery
  Sleep quality is assessed with Pittsburgh Sleep Quality Index (PSQI).

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Xuan Liu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (6):
- China (6):
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of JiNan University, Guangzhou, Guangdong
  - The Eighth Affliated Hospital of Southern Medical Universily, Guangzhou, Guangdong
  - Ganzhou People's Hospital, Ganzhou, Jiangxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh ES, Fong TG, Hshieh TT, Inouye SK. Delirium in Older Persons: Advances in Diagnosis and Treatment. JAMA. 2017 Sep 26;318(12):1161-1174. doi: 10.1001/jama.2017.12067. PMID 28973626
- [Background] Rudolph JL, Marcantonio ER. Review articles: postoperative delirium: acute change with long-term implications. Anesth Analg. 2011 May;112(5):1202-11. doi: 10.1213/ANE.0b013e3182147f6d. Epub 2011 Apr 7. PMID 21474660
- [Background] Lindroth H, Bratzke L, Purvis S, Brown R, Coburn M, Mrkobrada M, Chan MTV, Davis DHJ, Pandharipande P, Carlsson CM, Sanders RD. Systematic review of prediction models for delirium in the older adult inpatient. BMJ Open. 2018 Apr 28;8(4):e019223. doi: 10.1136/bmjopen-2017-019223. PMID 29705752
- [Background] Balas MC, Happ MB, Yang W, Chelluri L, Richmond T. Outcomes Associated With Delirium in Older Patients in Surgical ICUs. Chest. 2009 Jan;135(1):18-25. doi: 10.1378/chest.08-1456. Epub 2008 Nov 18. PMID 19017895
- [Background] Salluh JI, Wang H, Schneider EB, Nagaraja N, Yenokyan G, Damluji A, Serafim RB, Stevens RD. Outcome of delirium in critically ill patients: systematic review and meta-analysis. BMJ. 2015 Jun 3;350:h2538. doi: 10.1136/bmj.h2538. PMID 26041151
- [Background] Moskowitz EE, Overbey DM, Jones TS, Jones EL, Arcomano TR, Moore JT, Robinson TN. Post-operative delirium is associated with increased 5-year mortality. Am J Surg. 2017 Dec;214(6):1036-1038. doi: 10.1016/j.amjsurg.2017.08.034. Epub 2017 Sep 20. PMID 28947274
- [Background] Crocker E, Beggs T, Hassan A, Denault A, Lamarche Y, Bagshaw S, Elmi-Sarabi M, Hiebert B, Macdonald K, Giles-Smith L, Tangri N, Arora RC. Long-Term Effects of Postoperative Delirium in Patients Undergoing Cardiac Operation: A Systematic Review. Ann Thorac Surg. 2016 Oct;102(4):1391-9. doi: 10.1016/j.athoracsur.2016.04.071. Epub 2016 Jun 22. PMID 27344279
- [Background] Maclullich AM, Ferguson KJ, Miller T, de Rooij SE, Cunningham C. Unravelling the pathophysiology of delirium: a focus on the role of aberrant stress responses. J Psychosom Res. 2008 Sep;65(3):229-38. doi: 10.1016/j.jpsychores.2008.05.019. PMID 18707945
- [Background] Zhao J, Zhang R, Wang W, Jiang S, Liang H, Guo C, Qi J, Zeng H, Song H. Low-dose ketamine inhibits neuronal apoptosis and neuroinflammation in PC12 cells via alpha7nAChR mediated TLR4/MAPK/NF-kappaB signaling pathway. Int Immunopharmacol. 2023 Apr;117:109880. doi: 10.1016/j.intimp.2023.109880. Epub 2023 Feb 27. PMID 36842233
- [Background] Chen M, Han Y, Que B, Zhou R, Gan J, Dong X. Prophylactic Effects of Sub-anesthesia Ketamine on Cognitive Decline, Neuroinflammation, and Oxidative Stress in Elderly Mice. Am J Alzheimers Dis Other Demen. 2022 Jan-Dec;37:15333175221141531. doi: 10.1177/15333175221141531. PMID 36474365
- [Background] Faisal H, Qamar F, Hsu ES, Xu J, Lai EC, Wong ST, Masud FN. Prevalence of Delirium After Abdominal Surgery and Association With Ketamine: A Retrospective, Propensity-Matched Cohort Study. Crit Care Explor. 2024 Jan 11;6(1):e1032. doi: 10.1097/CCE.0000000000001032. eCollection 2024 Jan. PMID 38222873
- [Background] Hudetz JA, Patterson KM, Iqbal Z, Gandhi SD, Byrne AJ, Hudetz AG, Warltier DC, Pagel PS. Ketamine attenuates delirium after cardiac surgery with cardiopulmonary bypass. J Cardiothorac Vasc Anesth. 2009 Oct;23(5):651-7. doi: 10.1053/j.jvca.2008.12.021. Epub 2009 Feb 23. PMID 19231245
- [Background] Avidan MS, Maybrier HR, Abdallah AB, Jacobsohn E, Vlisides PE, Pryor KO, Veselis RA, Grocott HP, Emmert DA, Rogers EM, Downey RJ, Yulico H, Noh GJ, Lee YH, Waszynski CM, Arya VK, Pagel PS, Hudetz JA, Muench MR, Fritz BA, Waberski W, Inouye SK, Mashour GA; PODCAST Research Group. Intraoperative ketamine for prevention of postoperative delirium or pain after major surgery in older adults: an international, multicentre, double-blind, randomised clinical trial. Lancet. 2017 Jul 15;390(10091):267-275. doi: 10.1016/S0140-6736(17)31467-8. Epub 2017 May 30. PMID 28576285
- [Background] Fellous S, Dubost B, Cambriel A, Bonnet MP, Verdonk F. Perioperative ketamine administration to prevent delirium and neurocognitive disorders after surgery: a systematic review and meta-analysis. Int J Surg. 2023 Nov 1;109(11):3555-3565. doi: 10.1097/JS9.0000000000000619. PMID 37526094
- [Background] Pfenninger EG, Durieux ME, Himmelseher S. Cognitive impairment after small-dose ketamine isomers in comparison to equianalgesic racemic ketamine in human volunteers. Anesthesiology. 2002 Feb;96(2):357-66. doi: 10.1097/00000542-200202000-00022. PMID 11818769
- [Background] Xiong X, Shao Y, Chen D, Chen B, Lan X, Shi J. Effect of Esketamine on Postoperative Delirium in Patients Undergoing Cardiac Valve Replacement with Cardiopulmonary Bypass: A Randomized Controlled Trial. Anesth Analg. 2024 Oct 1;139(4):743-753. doi: 10.1213/ANE.0000000000006925. Epub 2024 Mar 6. PMID 38446699
- [Background] Ma J, Wang F, Wang J, Wang P, Dou X, Yao S, Lin Y. The Effect of Low-Dose Esketamine on Postoperative Neurocognitive Dysfunction in Elderly Patients Undergoing General Anesthesia for Gastrointestinal Tumors: A Randomized Controlled Trial. Drug Des Devel Ther. 2023 Jun 29;17:1945-1957. doi: 10.2147/DDDT.S406568. eCollection 2023. PMID 37408867
- [Background] Liu J, Wang T, Song J, Cao L. Effect of esketamine on postoperative analgesia and postoperative delirium in elderly patients undergoing gastrointestinal surgery. BMC Anesthesiol. 2024 Feb 1;24(1):46. doi: 10.1186/s12871-024-02424-w. PMID 38302882
- [Background] Bornemann-Cimenti H, Wejbora M, Michaeli K, Edler A, Sandner-Kiesling A. The effects of minimal-dose versus low-dose S-ketamine on opioid consumption, hyperalgesia, and postoperative delirium: a triple-blinded, randomized, active- and placebo-controlled clinical trial. Minerva Anestesiol. 2016 Oct;82(10):1069-1076. Epub 2016 Jun 21. PMID 27327855
- [Background] Lin X, Liu X, Huang H, Xu X, Zhang T, Gao J. Esketamine and neurocognitive disorders in adult surgical patients: a meta-analysis. BMC Anesthesiol. 2024 Dec 5;24(1):448. doi: 10.1186/s12871-024-02803-3. PMID 39639216
- [Background] Zhang W, Wang D, Li S, Chen Y, Bi C. Effect of esketamine on postoperative delirium in general anesthesia patients undergoing elective surgery: a meta-analysis of randomized controlled trials. BMC Anesthesiol. 2024 Nov 28;24(1):442. doi: 10.1186/s12871-024-02833-x. PMID 39609668
- [Background] Zhang Y, Chen R, Tang S, Sun T, Yu Y, Shi R, Wang K, Zeng Z, Liu X, Meng Q, Xia Z. Diurnal variation of postoperative delirium in elderly patients undergoing esketamine anesthesia for elective noncardiac surgery: a randomized clinical trial. Int J Surg. 2024 Sep 1;110(9):5496-5504. doi: 10.1097/JS9.0000000000001642. PMID 39275772
- [Background] Huang C, Yang R, Xie X, Dai H, Pan L. Effect of small dose esketamine on perioperative neurocognitive disorder and postoperative depressive symptoms in elderly patients undergoing major elective noncardiac surgery for malignant tumors: A randomized clinical trial. Medicine (Baltimore). 2024 Oct 18;103(42):e40028. doi: 10.1097/MD.0000000000040028. PMID 39432604
- [Background] Ma CB, Zhang CY, Gou CL, Liang ZH, Zhang JX, Xing F, Yuan JJ, Wei X, Zhang YB, Wang ZY. Effect of Low-Dose Esketamine on Postoperative Delirium in Elderly Patients Undergoing Total Hip or Knee Arthroplasty: A Randomized Controlled Trial. Drug Des Devel Ther. 2024 Nov 26;18:5409-5421. doi: 10.2147/DDDT.S477342. eCollection 2024. PMID 39624771
- [Background] Ormseth CH, LaHue SC, Oldham MA, Josephson SA, Whitaker E, Douglas VC. Predisposing and Precipitating Factors Associated With Delirium: A Systematic Review. JAMA Netw Open. 2023 Jan 3;6(1):e2249950. doi: 10.1001/jamanetworkopen.2022.49950. PMID 36607634
- [Background] Schuetz P, Seres D, Lobo DN, Gomes F, Kaegi-Braun N, Stanga Z. Management of disease-related malnutrition for patients being treated in hospital. Lancet. 2021 Nov 20;398(10314):1927-1938. doi: 10.1016/S0140-6736(21)01451-3. Epub 2021 Oct 14. PMID 34656286
- [Background] Mori N, Maeda K, Fujimoto Y, Nonogaki T, Ishida Y, Ohta R, Shimizu A, Ueshima J, Nagano A, Fukushima R. Prognostic implications of the global leadership initiative on malnutrition criteria as a routine assessment modality for malnutrition in hospitalized patients at a university hospital. Clin Nutr. 2023 Feb;42(2):166-172. doi: 10.1016/j.clnu.2022.12.008. Epub 2022 Dec 22. PMID 36586218
- [Background] GBD 2016 Alcohol Collaborators. Alcohol use and burden for 195 countries and territories, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2018 Sep 22;392(10152):1015-1035. doi: 10.1016/S0140-6736(18)31310-2. Epub 2018 Aug 23. PMID 30146330
- [Background] Cao SJ, Zhang Y, Zhang YX, Zhao W, Pan LH, Sun XD, Jia Z, Ouyang W, Ye QS, Zhang FX, Guo YQ, Ai YQ, Zhao BJ, Yu JB, Liu ZH, Yin N, Li XY, Ma JH, Li HJ, Wang MR, Sessler DI, Ma D, Wang DX; First Study of Perioperative Organ Protection (SPOP1) investigators. Delirium in older patients given propofol or sevoflurane anaesthesia for major cancer surgery: a multicentre randomised trial. Br J Anaesth. 2023 Aug;131(2):253-265. doi: 10.1016/j.bja.2023.04.024. Epub 2023 Jun 4. PMID 37474241
- [Background] Ghazaly HF, Hemaida TS, Zaher ZZ, Elkhodary OM, Hammad SS. A pre-anesthetic bolus of ketamine versus dexmedetomidine for prevention of postoperative delirium in elderly patients undergoing emergency surgery: a randomized, double-blinded, placebo-controlled study. BMC Anesthesiol. 2023 Dec 11;23(1):407. doi: 10.1186/s12871-023-02367-8. PMID 38082227
- [Background] Ren Q, Hua L, Zhou X, Cheng Y, Lu M, Zhang C, Guo J, Xu H. Effects of a Single Sub-Anesthetic Dose of Ketamine on Postoperative Emotional Responses and Inflammatory Factors in Colorectal Cancer Patients. Front Pharmacol. 2022 Apr 5;13:818822. doi: 10.3389/fphar.2022.818822. eCollection 2022. PMID 35479322